CLINICAL TRIAL: NCT06481826
Title: A Study to Evaluate Glofitamab as Single Agent in Chinese Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Glofitamab in Chinese Patients With R/R DLBCL
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Glofitamab-1
Record Dates: First submitted 2024-06-12; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — glofitamab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- treatment group: Glofitamab
  Interventions: Drug: Glofitamab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab given in standard dosage

SUMMARY:
This study will evaluate the safety and efficacy of glofitamab as a single agent in Chinese patients with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL) who have failed two or more lines of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed DLBCL
2. Participants must have relapsed or failed to respond to at least two lines of prior systemic therapy
3. Participants must have measurable disease

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Patient with known active infection, or reactivation of a latent infection
3. Patient with active autoimmune disease or immune deficiency
4. severe organ failure：LVEF<40%；DLCO<40%；eGFR<30ml/min；Bilirubin≥3ULN
5. Patients who are dependent on the sponsor, the investigator or the trial site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  Progression-free survival

SECONDARY OUTCOMES:
OS | 2 year
  overall survival
CR rate | 6 weeks, 18 weeks, 36 weeks
  complete response
ORR | 6 weeks, 18 weeks, 36 weeks
  overall response rate
DOR | 2 year
  duration of response
AE | 2 year
  Rate and type of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
the study protocol, statistical analysis plan, informed consent form, clinical study report would be available upon email request in 3 years after the closure of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years after the closure of the study
Access Criteria: upon email request

REFERENCES:
- [Background] Dickinson MJ, Carlo-Stella C, Morschhauser F, Bachy E, Corradini P, Iacoboni G, Khan C, Wrobel T, Offner F, Trneny M, Wu SJ, Cartron G, Hertzberg M, Sureda A, Perez-Callejo D, Lundberg L, Relf J, Dixon M, Clark E, Humphrey K, Hutchings M. Glofitamab for Relapsed or Refractory Diffuse Large B-Cell Lymphoma. N Engl J Med. 2022 Dec 15;387(24):2220-2231. doi: 10.1056/NEJMoa2206913. Epub 2022 Dec 11. PMID 36507690
- [Background] Birtas Atesoglu E, Gulbas Z, Uzay A, Ozcan M, Ozkalemkas F, Dal MS, Kalyon H, Akay OM, Deveci B, Bekoz H, Sevindik OG, Toptas T, Yilmaz F, Koyun D, Alkis N, Alacacioglu I, Sonmez M, Yavasoglu I, Tombak A, Mehtap O, Kurnaz F, Yuce OK, Karakus V, Turgut M, Kurekci DD, Ayer M, Keklik M, Buyuktas D, Ozbalak M, Ferhanoglu B. Glofitamab in relapsed/refractory diffuse large B-cell lymphoma: Real-world data. Hematol Oncol. 2023 Oct;41(4):663-673. doi: 10.1002/hon.3174. Epub 2023 May 22. PMID 37211991
- [Background] Song YQ, Zhang HL, Huang HQ, Zhang QY, Jing HM, Wang C, Wu C, Li DH, Dai Y, Humphrey K, Zhu J. Glofitamab monotherapy induces high complete response rates and manageable safety in Chinese patients with heavily pretreated relapsed or refractory diffuse large B-cell lymphoma. Haematologica. 2024 Apr 1;109(4):1269-1273. doi: 10.3324/haematol.2023.283802. No abstract available. PMID 37855035